CLINICAL TRIAL: NCT00269867
Title: A Placebo-Controlled, Double-Blinded, Randomized Clinical Trial of Anti-TNF Chimeric Monoclonal Antibody (cA2) in Patients With Active Rheumatoid Arthritis Despite Methotrexate Treatment
Brief Title: Infliximab Plus Methotrexate for the Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006259
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; infliximab; methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Matching placebo will be adminstered at Week 0, 2, 6 and every 4 weeks up to Week 54.
  Interventions: Drug: Placebo
- Infliximab 3 mg/kg every 8 weeks (Experimental): Infliximab 3 milligram per kilogram (mg/kg) will be administered as infusion at Week 0, 2, 6 and every 8 weeks up to Week 52.
  Interventions: Drug: Infliximab 3 mg/kg
- Infliximab 3 mg/kg every 4 weeks (Experimental): Infliximab 3 mg/kg will be administered as infusion at Week 0, 2, 6 and every 4 weeks up to Week 52.
  Interventions: Drug: Infliximab 3 mg/kg
- Infliximab 10 mg/kg every 8 weeks (Experimental): Infliximab 10 mg/kg will be administered as infusion at Week 0, 2, 6 and every 8 weeks up to Week 52.
  Interventions: Drug: Infliximab 10 mg/kg
- Infliximab 10 mg/kg every 4 weeks (Experimental): Infliximab 3 mg/kg will be administered as infusion at Week 0, 2, 6 and every 4 weeks up to Week 52.
  Interventions: Drug: Infliximab 10 mg/kg

INTERVENTIONS:
Drug: Placebo — Matching placebo will be adminstered at Week 0, 2, 6 and every 4 weeks up to Week 54.
  Arms: Placebo
Drug: Infliximab 3 mg/kg — Infliximab (anti-TNF chimeric monoclonal antibody [cA2]) 3 milligram per kilogram (mg/kg) will be administered as infusion at Week 0, 2, 6 and every 8 weeks or every 4 weeks up to Week 52.
  Other Names: anti-TNF chimeric monoclonal antibody (cA2)
  Arms: Infliximab 3 mg/kg every 4 weeks; Infliximab 3 mg/kg every 8 weeks
Drug: Infliximab 10 mg/kg — Infliximab (anti-TNF chimeric monoclonal antibody [cA2]) 3 milligram per kilogram (mg/kg) will be administered as infusion at Week 0, 2, 6 and every 8 weeks or every 4 weeks up to Week 52.
  Other Names: anti-TNF chimeric monoclonal antibody (cA2)
  Arms: Infliximab 10 mg/kg every 4 weeks; Infliximab 10 mg/kg every 8 weeks

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of infliximab (an anti-TNF chimeric monoclonal antibody [cA2]) in patients with active Rheumatoid Arthritis, despite methotrexate treatment.

DETAILED DESCRIPTION:
This is a placebo-controlled, double-blinded, randomized clinical study to evaluate the safety and effectiveness of infliximab in patients with active Rheumatoid Arthritis, despite methotrexate treatment. Infliximab is an anti-TNF chimeric monoclonal antibody (cA2). The primary measures of effectiveness include the change from baseline in American College of Rheumatology (ACR20) response at week 30, and the change in the modified van der Heijde Sharp Score. The ACR20 Responder Index a composite of clinical, laboratory, and functional measures and the van der Heijde-Sharp (vdH-S) scoring method is a method of rating structural damage in patients..

Patients will be treated with either infliximab or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active Rheumatoid Arthritis despite treatment with methotrexate
* Diagnosed with Rheumatoid Arthritis at least 6 months prior to screening
* Having active disease at the time of screening and pre-infusion as defined by having at least 6 or more swollen joints and 6 or more tender joints
* Using methotrexate for at least 3 months prior to study enrollment

Exclusion Criteria:

* Patients having any systemic inflammatory condition
* Having Lyme disease or a rheumatic disease other than Rheumatoid Arthritis
* Who have used Disease-Modifying Antirheumatic Drugs (DMARDs) other than methotrexate within 4 weeks prior to screening
* Who have used corticosteroids within 4 weeks prior to screening
* Having received previous administration of infliximab

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 1997-03; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in ACR20 response at week 30; Change in modified van der Heijde-Sharp Score | Baseline and Week 30

SECONDARY OUTCOMES:
safety | up to Week 54

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.

REFERENCES:
- [Result] Lipsky PE, van der Heijde DM, St Clair EW, Furst DE, Breedveld FC, Kalden JR, Smolen JS, Weisman M, Emery P, Feldmann M, Harriman GR, Maini RN; Anti-Tumor Necrosis Factor Trial in Rheumatoid Arthritis with Concomitant Therapy Study Group. Infliximab and methotrexate in the treatment of rheumatoid arthritis. Anti-Tumor Necrosis Factor Trial in Rheumatoid Arthritis with Concomitant Therapy Study Group. N Engl J Med. 2000 Nov 30;343(22):1594-602. doi: 10.1056/NEJM200011303432202. PMID 11096166
- [Derived] Mack ME, Hsia E, Aletaha D. Comparative Assessment of the Different American College of Rheumatology/European League Against Rheumatism Remission Definitions for Rheumatoid Arthritis for Their Use as Clinical Trial End Points. Arthritis Rheumatol. 2017 Mar;69(3):518-528. doi: 10.1002/art.39945. PMID 27696724